CLINICAL TRIAL: NCT04776993
Title: A Phase III, Randomized, Controlled, Open Label, no Profit, Single-center Intervention Study to Compare the Effect of a Conservative (Antithyroid Drugs) and an Ablative Approach (Radioiodine or Total Thyroidectomy) for the Treatment of Hyperthyroidism in Patients With Graves' Disease and Moderate-to-severe and Active Graves' Orbitopathy (GO) Treated With Intravenous Glucocorticoids (ABLAGO Study)
Brief Title: A Conservative vs an Ablative Approach for Treatment of Hyperthyroidism in Patients With Graves' Orbitopathy
Acronym: ABLAGO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Marinò Michele, Associate Professor, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABLAGO
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Graves' Orbitopathy
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Methimazole; Iodine-131; Thyroidectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methimazole (Experimental): Antithyroid drugs (at individualized dosage) for 72 weeks and a cumulative dose of 4.5 g of methylprednisolone divided into 12 weekly infusions
  Interventions: Drug: Methimazole
- Thyroid ablation (Active Comparator): Radioiodine therapy or total thyroidectomy (according to ultrasound thyroid volume) and a cumulative dose of 4.5 g of methylprednisolone divided into 12 weekly infusions
  Interventions: Procedure: Radioiodine or thyroidectomy

INTERVENTIONS:
Drug: Methimazole — Methimazole for 72 weeks
  Other Names: MMI
  Arms: Methimazole
Procedure: Radioiodine or thyroidectomy — Treatment with radioiodine or with thyroidectomy
  Other Names: Thyroid ablation
  Arms: Thyroid ablation

SUMMARY:
Graves' disease (GD) is the most frequent cause of hyperthyroidism in iodine sufficient countries and Graves' orbitopathy (GO) is its most common extrathyroidal manifestation. Restoration and maintenance of euthyroidism are imperative in Graves' disease patients with GO. The main treatment options for Graves' hyperthyroidism are antithyroid drugs, radioactive iodine (RAI), and surgery. Whether one or the other therapy for Graves' hyperthyroidism offers the best protection against GO is not established. The study is aimed at comparing the effects of a conservative approach (antithyroid drugs, ATDs, experimental arm) vs an ablative approach (radioiodine or total thyroidectomy) of thyroid treatment on the overall outcome of GO in patients with GD and moderate-to-severe and active GO treated with intravenous glucocorticoids.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing and capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
2. A diagnosis of Graves' disease based on the presence of hyperthyroidism associated with detectable anti-thyrotropic hormone (TSH) receptor autoantibodies (TRAb). Patients must be euthyroid under control on stable medical regimen and every effort will be made to maintain the euthyroid status for the entire duration of the clinical trial.
3. Duration of Graves' disease shorter than 18 months
4. A moderate-to-severe GO, defined as the presence of at least one of the following criteria in the most affected eye: an exophthalmos ≥2 mm compared with normal values for sex and race; presence of inconstant to constant diplopia; a lid retraction ≥2 mm
5. Active GO: CAS ≥ 3 out of 7 points in the most affected eye. Taking into account severity (moderate-to-severe) and activity (CAS ≥ 3/7) of GO, patients are eligible for methylprednisolone treatment according to clinical practice.
6. Duration of GO shorter than 18 months
7. Male and female patients of age 18-75 years
8. Compliant patient, regular follow-up possible

Exclusion Criteria:

1. Optic neuropathy
2. Previous therapy for Graves' disease with radioiodine or thyroidectomy
3. Corticosteroids or other immunosuppressive treatment for GO or other reasons in the last 3 months.
4. Previous surgical treatment and/or radiotherapy for GO
5. Contraindications to GC: hypersensitivity to the active substance or to any of the excipients; uncontrolled hypertension, uncontrolled diabetes; history of peptic ulcer; urinary infections, glaucoma, systemic fungal infections, systemic infections unless appropriate therapy is employed, idiopathic thrombocytopenic purpura, cerebral edema associated with malaria.
6. Use of medications interfering with GC or increasing the risk of GC-related adverse events (see prohibited therapies)
7. Acute or chronic liver disease
8. Contraindications to ATD: hypersensitivity to the active substance or to any of the excipients; breastfeeding
9. Women of childbearing potential (WOCBP, namely not in menopause or in menopause since less than two years; in all other instances women will be considered as non-WOCBP) and men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year (as indicated in Appendix) for at least 6 and 7,5 months, respectively, after the last dose of the investigational drug (see also 2014_09_HMA_CTFG_Contraception.pdf, namely the "2014 CTFG Reccommendtions related to contraception and pregnancy testing in clinical trials")
10. Contraindications of any kind to perform thyroidectomy
11. Mental illness that prevent patients from comprehensive, written informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall GO outcome | 24 weeks
  Improvement is defined as change in two of the following outcome measures in at least one eye, without deterioration in any of the same measures in both eyes (compared to baseline):
  * Improvement in CAS by at least 2 points
  * Improvement in exophthalmos by at least 2 mm (Hertel exophthalmometer)
  * Improvement in lid aperture by at least 2 mm
  * Improvement in diplopia (disappearance or change in the degree)
  * Improvement of visual acuity by at least 0.2/1
  Patients meeting the improvement criteria will be considered as "responders". All other patients will be considered as "non-responders".

SECONDARY OUTCOMES:
Overall GO outcome | 48 weeks
  Improvement is defined as change in two of the following outcome measures in at least one eye, without deterioration in any of the same measures in both eyes (compared to baseline):
  * Improvement in CAS by at least 2 points
  * Improvement in exophthalmos by at least 2 mm (Hertel exophthalmometer)
  * Improvement in lid aperture by at least 2 mm
  * Improvement in diplopia (disappearance or change in the degree)
  * Improvement of visual acuity by at least 0.2/1
  Patients meeting the improvement criteria will be considered as "responders". All other patients will be considered as "non-responders".
Overall GO outcome | 72 weeks
  Improvement is defined as change in two of the following outcome measures in at least one eye, without deterioration in any of the same measures in both eyes (compared to baseline):
  * Improvement in CAS by at least 2 points
  * Improvement in exophthalmos by at least 2 mm (Hertel exophthalmometer)
  * Improvement in lid aperture by at least 2 mm
  * Improvement in diplopia (disappearance or change in the degree)
  * Improvement of visual acuity by at least 0.2/1
  Patients meeting the improvement criteria will be considered as "responders". All other patients will be considered as "non-responders".
Response of individual GO parameters: proptosis, CAS, eyelid width, diplopia, and visual acuity | 24, 48 and 72 weeks
  Improvement is defined as change in each of the following outcome measures in at least one eye, without deterioration in both eyes (compared to baseline):
  * Improvement in CAS by at least 2 points
  * Improvement in exophthalmos by at least 2 mm (Hertel exophthalmometer)
  * Improvement in lid aperture by at least 2 mm
  * Improvement in diplopia (disappearance or change in the degree)
  * Improvement of visual acuity by at least 0.2/1
  Patients meeting the improvement criteria will be considered as "responders". All other patients will be considered as "non-responders".
Quality of life questionnaire | 24, 48 and 72 weeks
  Comparison of a disease specific quality of life questionnaire (GO-QoL) at 24, 48 and 72 weeks. Positive response: an improvement in the questionnaire by at least 6/48 points. The GO-QoL contains 8 questions on visual functioning and 8 questions on appearance. The minimal clinically important difference in scores is ≥ 10 points for invasive therapies, but a change of 6 is already perceived by patients as beneficial and is associated with an important change in daily functioning. The GO-QoL is well validated, widely used, and available in eight languages. The GO-QoL is recommended as an independent outcome measure in randomized clinical trials24.

CONTACTS AND LOCATIONS:
Locations (1):
- Endocrinology Unit II, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: No